CLINICAL TRIAL: NCT04842968
Title: The Impact of ex Vivo Intra-arterial Methylene Blue Injection on Nodal Staging Accuracy and Survival in Colorectal Cancer.
Brief Title: Ex Vivo Intraarterial Methylene Blue Injection Improve Nodal Staging Accuracy in Colorectal Cancer
Acronym: MB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Borbala Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IV/3228/2021-EKU
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2021-04

CONDITIONS: Lymph Node Metastases; Colorectal Cancer
Keywords: colorectal; cancer; lymph; node; metastasis; methylene-blue
MeSH Terms: conditions — Lymphatic Metastasis; Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Methylene Blue

STUDY DESIGN:
Intervention Model Description: Five to six years ago specimens from a total fo 200 consecutive colorectal cancer resection cases were randomized into two groups: 1. main supplying artery was cannulated and injected with methylene blue solution, 2. no intervention, routine specimen handling.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue (Experimental): Methylene blue solution (50 mg in 30 ml of saline solution) was injected in the cannulated main supplying artery of the freshly removed specimen, ex vivo. Colorectal specimen was then processed in the routine pathological work-up way.
  Interventions: Other: Methylene blue injection
- Control (No Intervention): Colorectal specimens were processed in the routine pathological work-up way.

INTERVENTIONS:
Other: Methylene blue injection — Methylene blue solution is injected ex vivo in the main supplying artery trunk of the freshly removed colorectal specimen. (50 mg in 30 ml saline)
  Arms: Methylene blue

SUMMARY:
Nodal staging holds both important prognostic and predictive value at colorectal cancer. Regional lymph nodes are located close to the primary tumor in the mesocolon / mesorectum. Current pathology and oncology standards require a separate examination of at least 12 lymph nodes each case to fulfill staging "accuracy" criteria.

In order to reach this number of lymph nodes, a precise surgical technique (total mesorectal excision or complete mesocolic excision), as well as a thorough pathological specimen work-up is needed.

The aim of the study is to investigate, if ex vivo intra-arterial methylene blue injection by the surgeon can help improving nodal harvesting effectivity of the pathologist, hence leading to a better staging and hopefully even to a better outcome in the long run.

In 2014-2015 two surgical centers randomised resected colorectal specimens in 1:1 ratio to methylene-blue injection arm and control (no injection) arm in a total of 200 consecutive cases. Both pathologic and oncologic treatment were led regardless of the injection, reports were just routinely saved in the routine medical documentation.

This retrospective study is designed to recall patient-related, surgery-related factors, as well as pathology reports including nodal staging from the medical databases. The investigators aim to find correlation between methylene blue "staining" and lymph node yield. In addition, the investigators plan to crossmatch methylene blue injection, as a process, with long term survival of the patients.

DETAILED DESCRIPTION:
Background:

Colorectal Cancer is the second most common cause of death in Hungary. The most important prognostic and predictive factor of colorectal cancer is the stage of disease at the time of diagnosis. Precise staging, especially nodal staging is highly important for correct planning of oncotherapy, i.e. adjuvant chemotherapy. Nodal staging relies on the proper surgical removal of mesocolon/mesorectum belonging to the the affected colorectal segment, as well as on the thorough pathology work-up of the specimen.

Current quality standards require examination of a minimum of 12 lymph nodes in order to reliably report N0 stage.

Methylene-blue injection into the main supplying artery of the removed specimen is one of the simplest and most effective techniques described to aid pathologist in lymph node harvesting.

Technique of methylene blue injection:

First of all, surgeon need to en block remove the affected colorectal segment with its mesecolon/mesorectum. Then the surgeon isolates the main supplying artery and cannulated it with an appropriate-size canula.

Methylene blue solution (50 mg methylene blue diluted in in 30 ml saline) is prepared and injected into the freshly removed specimen via the canula until the blue solution appears on the cut edges of the specimen.

The specimen can be processed in a routine way (placed in 4% formaldehyde).

Aim of the study:

The aim is to investigate if the well described and in Western-European healthcare systems well tested technique (Methylene blue injection) can be effectively adapted in an overwhelmed, busy Eastern-European healthcare environment. (Other techniques, including pathology assistant are not affordable in this area.) Apart form testing diagnostic accuracy of the pathologist on specimens with and without methylene blue injection, the investigators would like to assess a potential survival benefit of the suspected improvement of staging effectivity.

Timing of the study:

Over a 20-month period of 2014 and 2015 two surgical centers in Hungary randomised their elective colorectal resection cases into interventional and control arms. Randomisation was performed with a 1:1 ratio at each site on 100-100 consecutive cases.

Further pathology work-up and reporting has been routinely performed without any specific effect on oncology follow-up or treatment. No specific data collection has been performed after the intervention.

This study aims to retrospectively select the 100-100 (total of 200) consecutive colorectal resection cases of the given time frame from the official hospital medical recording systems.

Pathology reports and other relevant patient clinical records will be collected and statistically assessed.

Ethical approval was requested and gained from the Medical Research Council, Hungary, for the retrospective analysis of patient data.

Statistical analysis:

Power analysis was performed to get the sufficient number of cases (200 cases in total).

Case Report Form The retrospectively included cases will be listed in a specific database on a safe medical server. Anthropometric, disease-specific, operation-specific and pathology report details will be extracted out of the official patient documentation system.

Patients will be included according to the known interventional interval and the operation type (elective colorectal resection). Cases in the database will be anonymized. No patient-identifying data will be recorded or given to the assessor of the study (statistician).

ELIGIBILITY:
Inclusion Criteria:

* Elective operation.
* Colon or rectum resection performed.
* Malignant colorectal condition.
* Curative intent.

Exclusion Criteria:

* Acute surgery performed
* Final histology: benign
* No other pathologic method (apart form Methylene Blue injection) used to improve lymph node yield

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Total number of lymph nodes | Within 4 weeks after operation (at pathology work-up)
  Total number of lymph nodes examined by pathologist
Positive lymph nodes | Within 4 weeks after operation (at pathology work-up)
  Number of positive lymph nodes found by pathologist
Nodal staging accuracy | Within 4 weeks after operation (at pathology work-up)
  Minimum Nr of 12 lymph nodes examined if reported N stage is N0, or positive lymph node=s) found
At least 12 lymph nodes harvested | Within 4 weeks after operation (at pathology work-up)
  Minimum Nr of 12 lymph nodes examined by pathologist

SECONDARY OUTCOMES:
Overall survival | 5 years (60 months) after operation
  Overall survival after operation (in months)

CONTACTS AND LOCATIONS:
Overall Officials: Balazs Banky, PhD, Principal Investigator — St. Borbala Hospital
Locations (1):
- St. Borbala Hospital, Tatabánya, Hungary

IPD SHARING:
Plan to Share IPD: No